CLINICAL TRIAL: NCT01231958
Title: The Boston Puerto Rican Health Study: Center for Population Health and Health Disparities
Brief Title: Boston Puerto Rican Health Study
Acronym: BPRHS
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Lowell (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute on Aging (NIA) (NIH); Tufts University (Other); Northeastern University (Other)
Responsible Party: Principal Investigator, Katherine Tucker, Professor, University of Massachusetts, Lowell
Other Study IDs: P50HL105185 (NIH); P01AG023394 (NIH)
Record Dates: First submitted 2010-10-04; First posted 2010-11-01 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Risk Factor
Keywords: Puerto Rican; CVD; Hispanic; health disparities; allostatic load; diet
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, saliva
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: The Heart Healthy Initiative for Hispanic Adults (HIP) — This randomized controlled pilot intervention study will include 150 Hispanic adults (45-75y) in the Greater Boston area. Participants will be randomized to either the intervention or control group after completing their baseline interview. The intervention group will receive 6 months of weekly group educational sessions, Zumba fitness classes and interactions with an embodied computer agent (ECA). The fitness classes and interactions with the ECA will continue for the second 6 months of the 1 year intervention. Intervention activities will occur at community centers in the greater Boston area. Control participants will receive standard of care for the first 6 months and will be offered the full intervention (weekly group educational sessions, Zumba fitness classes and interactions with the ECA) for the second 6 months of the study. Participants will complete an interview and blood draw at baseline, 6 months, and 12 months.

SUMMARY:
The investigators long-term goal is to understand the complex interactions of diet and other behavioral and environmental factors, genetics, and psychosocial stress on the high and apparently increasing prevalence of cardiovascular disease (CVD) risk factors in Puerto Rican adults.

DETAILED DESCRIPTION:
Puerto Rican adults living on the mainland US have documented health disparities; however, little research has been conducted with this second largest Hispanic subgroup. Our long-term goal is to understand the complex interactions of diet and other behavioral and environmental factors, genetics, and psychosocial stress on the high and apparently increasing prevalence of cardiovascular disease (CVD) risk factors in Puerto Rican adults. As this group is rapidly growing, understanding the reasons for this risk is of great importance. Our initial funding period for the Boston Puerto Rican Center for Population Health and Health Disparities (BPR-CPHHD, 2003-08) focused on the role of stress on physical disability and cognitive decline, through physiological dysregulation or "allostatic load." During that investigation, it became clear that risk factors for CVD were highly prevalent. These findings are in contrast to the commonly held belief that there is a Hispanic paradox--lower heart disease and mortality despite greater poverty. Importantly, the Puerto Rican population differs considerably in ancestral genetic history and in exposures to known risk factors from other Hispanic groups. They have unique dietary intake patterns, as well as social, cultural and environmental structures that contribute and affect reaction to stressors. During our initial funding period, we successfully assembled a cohort of 1500 Puerto Rican adults, aged 45-75 years at baseline, and completed two-year follow-up interviews on more than 1250 participants. As this population is aging and growing rapidly, the high prevalence and apparent cohort effect of increased heart disease risk factors suggest that 1) this population has serious health disparities in heart disease risk factors and 2) heart disease will become an even greater problem for this group in the near future. Our overall aim for this renewal is, therefore, to extend follow-up and to measure and analyze relevant characteristics and CVD risk factors, and to add additional contextual and outcome measures for CVD risk in this established cohort of Puerto Rican adults, so that we may better understand the dynamics of these disparities. Our model follows the transdisciplinary "cells to society" concept developed jointly with our partner CPHHDs during the initial funding period, with consideration of genetic variation in relation to longitudinal change in allostatic load and biochemical indicators of risk; with additional focus on social networks, neighborhood characteristics (physical space and access to food) and environment (air pollution) factors as social determinants of health. Finally, using community based participatory techniques, we will implement and test a multidimensional intervention that focuses on diet and exercise, but that also fully considers the social and physical environment to ensure success. With participation of our community partners, and the support of our administrative, biostatistics and laboratory cores, our team is efficiently poised to make significant contributions to understanding the factors that contribute to the apparent growing threat of heart disease in this highly disadvantaged group-while providing insights that may be useful to other vulnerable groups. The continuation of our cohort, with its rich constellation of measures, will allow us to unravel some of the complex etiologic interactions which contribute to CVD risk, so that effective interventions may be implemented. To date, we have completed approximately 840 5-year follow-up interviews.

ELIGIBILITY:
Inclusion Criteria:

* self-identified Puerto Rican decent
* aged 45-75 at baseline
* able to answer questions in English or Spanish
* living in the Boston, MA metropolitan area

Exclusion Criteria:

* unable to answer questions due to serious health conditions
* plan to move away from the area within two years
* Mini Mental State Examination (MMSE) score </=10

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Puerto Ricans older adults, aged 45-75 years, living in the Boston area.
Sampling Method: Non-Probability Sample
Enrollment: 1650 (Actual)
Dates: Start 2004-06; Primary Completion 2009-10 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Cardiovascular disease risk | 5 years

SECONDARY OUTCOMES:
10-year risk of Coronary Heart Disease (CHD) | 5 years
  10-year risk of CHD will be assessed using the Framingham Risk Score

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L. Tucker, PhD, Principal Investigator — University of Massachusetts, Lowell
Locations (3):
- United States (3):
  - Tufts University, Boston, Massachusetts
  - Northeastern University, Boston, Massachusetts
  - University of Massachusetts Lowell, Lowell, Massachusetts

REFERENCES:
- [Background] Warnecke RB, Oh A, Breen N, Gehlert S, Paskett E, Tucker KL, Lurie N, Rebbeck T, Goodwin J, Flack J, Srinivasan S, Kerner J, Heurtin-Roberts S, Abeles R, Tyson FL, Patmios G, Hiatt RA. Approaching health disparities from a population perspective: the National Institutes of Health Centers for Population Health and Health Disparities. Am J Public Health. 2008 Sep;98(9):1608-15. doi: 10.2105/AJPH.2006.102525. Epub 2008 Jul 16. PMID 18633099
- [Background] Paskett ED, Reeves KW, McLaughlin JM, Katz ML, McAlearney AS, Ruffin MT, Halbert CH, Merete C, Davis F, Gehlert S. Recruitment of minority and underserved populations in the United States: the Centers for Population Health and Health Disparities experience. Contemp Clin Trials. 2008 Nov;29(6):847-61. doi: 10.1016/j.cct.2008.07.006. Epub 2008 Jul 31. PMID 18721901
- [Background] Orho-Melander M, Melander O, Guiducci C, Perez-Martinez P, Corella D, Roos C, Tewhey R, Rieder MJ, Hall J, Abecasis G, Tai ES, Welch C, Arnett DK, Lyssenko V, Lindholm E, Saxena R, de Bakker PI, Burtt N, Voight BF, Hirschhorn JN, Tucker KL, Hedner T, Tuomi T, Isomaa B, Eriksson KF, Taskinen MR, Wahlstrand B, Hughes TE, Parnell LD, Lai CQ, Berglund G, Peltonen L, Vartiainen E, Jousilahti P, Havulinna AS, Salomaa V, Nilsson P, Groop L, Altshuler D, Ordovas JM, Kathiresan S. Common missense variant in the glucokinase regulatory protein gene is associated with increased plasma triglyceride and C-reactive protein but lower fasting glucose concentrations. Diabetes. 2008 Nov;57(11):3112-21. doi: 10.2337/db08-0516. Epub 2008 Aug 4. PMID 18678614
- [Background] Tucker KL, Mattei J, Noel SE, Collado BM, Mendez J, Nelson J, Griffith J, Ordovas JM, Falcon LM. The Boston Puerto Rican Health Study, a longitudinal cohort study on health disparities in Puerto Rican adults: challenges and opportunities. BMC Public Health. 2010 Mar 1;10:107. doi: 10.1186/1471-2458-10-107. PMID 20193082
- [Background] Fullerton SM, Anderson EE, Cowan K, Malen RC, Brugge D. Awareness of Federal Regulatory Mechanisms Relevant to Community-Engaged Research: Survey of Health Disparities-Oriented NIH-Funded Investigators. J Empir Res Hum Res Ethics. 2015 Feb;10(1):13-21. doi: 10.1177/1556264614561964. Epub 2014 Dec 10. PMID 25742662
- [Background] Cooper LA, Ortega AN, Ammerman AS, Buchwald D, Paskett ED, Powell LH, Thompson B, Tucker KL, Warnecke RB, McCarthy WJ, Viswanath KV, Henderson JA, Calhoun EA, Williams DR. Calling for a bold new vision of health disparities intervention research. Am J Public Health. 2015 Jul;105 Suppl 3(Suppl 3):S374-6. doi: 10.2105/AJPH.2014.302386. Epub 2015 Apr 23. No abstract available. PMID 25905830
- [Background] Glik D, Sharif MZ, Tucker KL, Tejada SA, Prelip ML, Ammerman AS, Keyserling TC, Torres SE, Pitts SJ. Community engagement to support cardiovascular disease prevention in disparities populations: three case studies. J Health Dispar Res Pract Apr 2016;9:71-87.
- [Result] Lai CQ, Tucker KL, Parnell LD, Adiconis X, Garcia-Bailo B, Griffith J, Meydani M, Ordovas JM. PPARGC1A variation associated with DNA damage, diabetes, and cardiovascular diseases: the Boston Puerto Rican Health Study. Diabetes. 2008 Apr;57(4):809-16. doi: 10.2337/db07-1238. Epub 2007 Dec 27. PMID 18162502
- [Result] Smith CE, Tucker KL, Yiannakouris N, Garcia-Bailo B, Mattei J, Lai CQ, Parnell LD, Ordovas JM. Perilipin polymorphism interacts with dietary carbohydrates to modulate anthropometric traits in hispanics of Caribbean origin. J Nutr. 2008 Oct;138(10):1852-8. doi: 10.1093/jn/138.10.1852. PMID 18806092
- [Result] DeVos L, Chanson A, Liu Z, Ciappio ED, Parnell LD, Mason JB, Tucker KL, Crott JW. Associations between single nucleotide polymorphisms in folate uptake and metabolizing genes with blood folate, homocysteine, and DNA uracil concentrations. Am J Clin Nutr. 2008 Oct;88(4):1149-58. doi: 10.1093/ajcn/88.4.1149. PMID 18842806
- [Result] Junyent M, Tucker KL, Smith CE, Garcia-Rios A, Mattei J, Lai CQ, Parnell LD, Ordovas JM. The effects of ABCG5/G8 polymorphisms on plasma HDL cholesterol concentrations depend on smoking habit in the Boston Puerto Rican Health Study. J Lipid Res. 2009 Mar;50(3):565-573. doi: 10.1194/jlr.P800041-JLR200. Epub 2008 Nov 12. PMID 19005228
- [Result] Perez-Martinez P, Corella D, Shen J, Arnett DK, Yiannakouris N, Tai ES, Orho-Melander M, Tucker KL, Tsai M, Straka RJ, Province M, Kai CS, Perez-Jimenez F, Lai CQ, Lopez-Miranda J, Guillen M, Parnell LD, Borecki I, Kathiresan S, Ordovas JM. Association between glucokinase regulatory protein (GCKR) and apolipoprotein A5 (APOA5) gene polymorphisms and triacylglycerol concentrations in fasting, postprandial, and fenofibrate-treated states. Am J Clin Nutr. 2009 Jan;89(1):391-9. doi: 10.3945/ajcn.2008.26363. Epub 2008 Dec 3. PMID 19056598
- [Result] Lai CQ, Tucker KL, Choudhry S, Parnell LD, Mattei J, Garcia-Bailo B, Beckman K, Burchard EG, Ordovas JM. Population admixture associated with disease prevalence in the Boston Puerto Rican health study. Hum Genet. 2009 Mar;125(2):199-209. doi: 10.1007/s00439-008-0612-7. Epub 2008 Dec 24. PMID 19107526
- [Result] Lai CQ, Parnell LD, Arnett DK, Garcia-Bailo B, Tsai MY, Kabagambe EK, Straka RJ, Province MA, An P, Borecki IB, Tucker KL, Ordovas JM. WDTC1, the ortholog of Drosophila adipose gene, associates with human obesity, modulated by MUFA intake. Obesity (Silver Spring). 2009 Mar;17(3):593-600. doi: 10.1038/oby.2008.561. Epub 2008 Dec 18. PMID 19238144
- [Result] Gao X, Scott T, Falcon LM, Wilde PE, Tucker KL. Food insecurity and cognitive function in Puerto Rican adults. Am J Clin Nutr. 2009 Apr;89(4):1197-203. doi: 10.3945/ajcn.2008.26941. Epub 2009 Feb 18. PMID 19225117
- [Result] Chanson A, Parnell LD, Ciappio ED, Liu Z, Crott JW, Tucker KL, Mason JB. Polymorphisms in uracil-processing genes, but not one-carbon nutrients, are associated with altered DNA uracil concentrations in an urban Puerto Rican population. Am J Clin Nutr. 2009 Jun;89(6):1927-36. doi: 10.3945/ajcn.2009.27429. Epub 2009 Apr 29. PMID 19403629
- [Result] Smith CE, Tucker KL, Scott TM, Van Rompay M, Mattei J, Lai CQ, Parnell LD, Junyent M, Lee YC, Garcia-Bailo B, Ordovas JM. Apolipoprotein C3 polymorphisms, cognitive function and diabetes in Caribbean origin Hispanics. PLoS One. 2009;4(5):e5465. doi: 10.1371/journal.pone.0005465. Epub 2009 May 8. PMID 19424489
- [Result] Noel SE, Newby PK, Ordovas JM, Tucker KL. A traditional rice and beans pattern is associated with metabolic syndrome in Puerto Rican older adults. J Nutr. 2009 Jul;139(7):1360-7. doi: 10.3945/jn.109.105874. Epub 2009 May 20. PMID 19458029
- [Result] Mattei J, Parnell LD, Lai CQ, Garcia-Bailo B, Adiconis X, Shen J, Arnett D, Demissie S, Tucker KL, Ordovas JM. Disparities in allele frequencies and population differentiation for 101 disease-associated single nucleotide polymorphisms between Puerto Ricans and non-Hispanic whites. BMC Genet. 2009 Aug 14;10:45. doi: 10.1186/1471-2156-10-45. PMID 19682384
- [Result] Smith CE, Tucker KL, Lai CQ, Parnell LD, Lee YC, Ordovas JM. Apolipoprotein A5 and lipoprotein lipase interact to modulate anthropometric measures in Hispanics of Caribbean origin. Obesity (Silver Spring). 2010 Feb;18(2):327-32. doi: 10.1038/oby.2009.216. Epub 2009 Jul 23. PMID 19629056
- [Result] Junyent M, Tucker KL, Smith CE, Lane JM, Mattei J, Lai CQ, Parnell LD, Ordovas JM. The effects of ABCG5/G8 polymorphisms on HDL-cholesterol concentrations depend on ABCA1 genetic variants in the Boston Puerto Rican Health Study. Nutr Metab Cardiovasc Dis. 2010 Oct;20(8):558-66. doi: 10.1016/j.numecd.2009.05.005. Epub 2009 Aug 18. PMID 19692220
- [Result] Junyent M, Tucker KL, Shen J, Lee YC, Smith CE, Mattei J, Lai CQ, Parnell LD, Ordovas JM. A composite scoring of genotypes discriminates coronary heart disease risk beyond conventional risk factors in the Boston Puerto Rican Health Study. Nutr Metab Cardiovasc Dis. 2010 Mar;20(3):157-64. doi: 10.1016/j.numecd.2009.03.016. Epub 2009 Jun 5. PMID 19501493
- [Result] Mattei J, Demissie S, Tucker KL, Ordovas JM. Apolipoprotein A5 polymorphisms interact with total dietary fat intake in association with markers of metabolic syndrome in Puerto Rican older adults. J Nutr. 2009 Dec;139(12):2301-8. doi: 10.3945/jn.109.109900. Epub 2009 Oct 14. PMID 19828688
- [Result] Falcon LM, Todorova I, Tucker K. Social support, life events, and psychological distress among the Puerto Rican population in the Boston area of the United States. Aging Ment Health. 2009 Nov;13(6):863-73. doi: 10.1080/13607860903046552. PMID 19888706
- [Result] Shen J, Lai CQ, Mattei J, Ordovas JM, Tucker KL. Association of vitamin B-6 status with inflammation, oxidative stress, and chronic inflammatory conditions: the Boston Puerto Rican Health Study. Am J Clin Nutr. 2010 Feb;91(2):337-42. doi: 10.3945/ajcn.2009.28571. Epub 2009 Dec 2. PMID 19955400
- [Result] Corella D, Peloso G, Arnett DK, Demissie S, Cupples LA, Tucker K, Lai CQ, Parnell LD, Coltell O, Lee YC, Ordovas JM. APOA2, dietary fat, and body mass index: replication of a gene-diet interaction in 3 independent populations. Arch Intern Med. 2009 Nov 9;169(20):1897-906. doi: 10.1001/archinternmed.2009.343. PMID 19901143
- [Result] Rioux CL, Tucker KL, Mwamburi M, Gute DM, Cohen SA, Brugge D. Residential traffic exposure, pulse pressure, and C-reactive protein: consistency and contrast among exposure characterization methods. Environ Health Perspect. 2010 Jun;118(6):803-11. doi: 10.1289/ehp.0901182. Epub 2010 Feb 2. PMID 20123638
- [Result] Henkin S, Tucker KL, Gao X, Falcon LM, Qawi I, Brugge D. Association of depression, psycho-social stress and acculturation with respiratory disease among Puerto Rican adults in Massachusetts. J Immigr Minor Health. 2011 Apr;13(2):214-23. doi: 10.1007/s10903-009-9307-y. PMID 20012203
- [Result] Noel SE, Lai CQ, Mattei J, Parnell LD, Ordovas JM, Tucker KL. Variants of the CD36 gene and metabolic syndrome in Boston Puerto Rican adults. Atherosclerosis. 2010 Jul;211(1):210-5. doi: 10.1016/j.atherosclerosis.2010.02.009. Epub 2010 Feb 18. PMID 20223461
- [Result] Mattei J, Demissie S, Falcon LM, Ordovas JM, Tucker K. Allostatic load is associated with chronic conditions in the Boston Puerto Rican Health Study. Soc Sci Med. 2010 Jun;70(12):1988-1996. doi: 10.1016/j.socscimed.2010.02.024. Epub 2010 Mar 15. PMID 20381934
- [Result] Castaneda-Sceppa C, Price LL, Noel SE, Bassett Midle J, Falcon LM, Tucker KL. Physical function and health status in aging Puerto Rican adults: the Boston Puerto Rican Health Study. J Aging Health. 2010 Aug;22(5):653-72. doi: 10.1177/0898264310366738. Epub 2010 May 21. PMID 20495158
- [Result] Noel SE, Newby PK, Ordovas JM, Tucker KL. Adherence to an (n-3) fatty acid/fish intake pattern is inversely associated with metabolic syndrome among Puerto Rican adults in the Greater Boston area. J Nutr. 2010 Oct;140(10):1846-54. doi: 10.3945/jn.110.124297. Epub 2010 Aug 11. PMID 20702744
- [Result] Gao X, Lai CQ, Scott T, Shen J, Cai T, Ordovas JM, Tucker KL. Urinary 8-hydroxy-2-deoxyguanosine and cognitive function in Puerto Rican adults. Am J Epidemiol. 2010 Aug 1;172(3):271-8. doi: 10.1093/aje/kwq136. Epub 2010 Jul 9. PMID 20621990
- [Result] Todorova IL, Falcon LM, Lincoln AK, Price LL. Perceived discrimination, psychological distress and health. Sociol Health Illn. 2010 Sep;32(6):843-61. doi: 10.1111/j.1467-9566.2010.01257.x. Epub 2010 Jul 23. PMID 20649891
- [Result] Ye X, Maras JE, Bakun PJ, Tucker KL. Dietary intake of vitamin B-6, plasma pyridoxal 5'-phosphate, and homocysteine in Puerto Rican adults. J Am Diet Assoc. 2010 Nov;110(11):1660-8. doi: 10.1016/j.jada.2010.08.006. PMID 21034879
- [Result] Lai CQ, Parnell LD, Troen AM, Shen J, Caouette H, Warodomwichit D, Lee YC, Crott JW, Qiu WQ, Rosenberg IH, Tucker KL, Ordovas JM. MAT1A variants are associated with hypertension, stroke, and markers of DNA damage and are modulated by plasma vitamin B-6 and folate. Am J Clin Nutr. 2010 May;91(5):1377-86. doi: 10.3945/ajcn.2009.28923. Epub 2010 Mar 24. PMID 20335551
- [Result] Bhupathiraju SN, Tucker KL. Greater variety in fruit and vegetable intake is associated with lower inflammation in Puerto Rican adults. Am J Clin Nutr. 2011 Jan;93(1):37-46. doi: 10.3945/ajcn.2010.29913. Epub 2010 Nov 10. PMID 21068354
- [Result] Mattei J, Demissie S, Tucker KL, Ordovas JM. The APOA1/C3/A4/A5 cluster and markers of allostatic load in the Boston Puerto Rican Health Study. Nutr Metab Cardiovasc Dis. 2011 Nov;21(11):862-70. doi: 10.1016/j.numecd.2010.02.024. Epub 2010 Jul 31. PMID 20674306
- [Result] Laugero KD, Falcon LM, Tucker KL. Relationship between perceived stress and dietary and activity patterns in older adults participating in the Boston Puerto Rican Health Study. Appetite. 2011 Feb;56(1):194-204. doi: 10.1016/j.appet.2010.11.001. Epub 2010 Nov 9. PMID 21070827
- [Result] Rioux CL, Tucker KL, Brugge D, Gute DM, Mwamburi M. Traffic exposure in a population with high prevalence type 2 diabetes--do medications influence concentrations of C-reactive protein? Environ Pollut. 2011 Aug-Sep;159(8-9):2051-60. doi: 10.1016/j.envpol.2010.12.025. Epub 2011 Feb 2. PMID 21292365
- [Result] Huang T, Tucker KL, Lee YC, Crott JW, Parnell LD, Shen J, Smith CE, Ordovas JM, Li D, Lai CQ. Methylenetetrahydrofolate reductase variants associated with hypertension and cardiovascular disease interact with dietary polyunsaturated fatty acids to modulate plasma homocysteine in puerto rican adults. J Nutr. 2011 Apr 1;141(4):654-9. doi: 10.3945/jn.110.134353. Epub 2011 Jan 26. PMID 21270364
- [Result] Van Rompay MI, Castaneda-Sceppa C, McKeown NM, Ordovas JM, Tucker KL. Prevalence of cardiovascular disease risk factors among older Puerto Rican adults living in Massachusetts. J Immigr Minor Health. 2011 Oct;13(5):825-33. doi: 10.1007/s10903-011-9448-7. PMID 21298483
- [Result] Ye X, Lai CQ, Crott JW, Troen AM, Ordovas JM, Tucker KL. The folate hydrolase 1561C>T polymorphism is associated with depressive symptoms in Puerto Rican adults. Psychosom Med. 2011 Jun;73(5):385-92. doi: 10.1097/PSY.0b013e31821a1ab4. Epub 2011 May 19. PMID 21597034
- [Result] Huang T, Tucker KL, Lee YC, Crott JW, Parnell LD, Shen J, Smith CE, Ordovas JM, Li D, Lai CQ. Interactions between genetic variants of folate metabolism genes and lifestyle affect plasma homocysteine concentrations in the Boston Puerto Rican population. Public Health Nutr. 2011 Oct;14(10):1805-12. doi: 10.1017/S1368980011000140. Epub 2011 Feb 22. PMID 21338559
- [Result] Ye X, Gao X, Scott T, Tucker KL. Habitual sugar intake and cognitive function among middle-aged and older Puerto Ricans without diabetes. Br J Nutr. 2011 Nov;106(9):1423-32. doi: 10.1017/S0007114511001760. Epub 2011 Jun 1. PMID 21736803
- [Result] Bhupathiraju SN, Lichtenstein AH, Dawson-Hughes B, Tucker KL. Adherence index based on the AHA 2006 diet and lifestyle recommendations is associated with select cardiovascular disease risk factors in older Puerto Ricans. J Nutr. 2011 Mar;141(3):460-9. doi: 10.3945/jn.110.133603. Epub 2011 Jan 26. PMID 21270369
- [Result] Oxenkrug G, Tucker KL, Requintina P, Summergrad P. Neopterin, a Marker of Interferon-Gamma-Inducible Inflammation, Correlates with Pyridoxal-5'-Phosphate, Waist Circumference, HDL-Cholesterol, Insulin Resistance and Mortality Risk in Adult Boston Community Dwellers of Puerto Rican Origin. Am J Neuroprot Neuroregen. 2011 Jun;3(1):48-52. doi: 10.1166/ajnn.2011.1024. PMID 22308202
- [Result] Mattei J, Noel SE, Tucker KL. A meat, processed meat, and French fries dietary pattern is associated with high allostatic load in Puerto Rican older adults. J Am Diet Assoc. 2011 Oct;111(10):1498-506. doi: 10.1016/j.jada.2011.07.006. PMID 21963016
- [Result] Corella D, Arnett DK, Tucker KL, Kabagambe EK, Tsai M, Parnell LD, Lai CQ, Lee YC, Warodomwichit D, Hopkins PN, Ordovas JM. A high intake of saturated fatty acids strengthens the association between the fat mass and obesity-associated gene and BMI. J Nutr. 2011 Dec;141(12):2219-25. doi: 10.3945/jn.111.143826. Epub 2011 Nov 2. PMID 22049296
- [Result] Huang T, Tucker K, Lee Y, Crott J, Parnell L, Shen J, Smith C, Ordovas J, Li D, Lai C. MAT1A variants modulate the effect of dietary fatty acids on plasma homocysteine concentrations. Nutr Metab Cardiovasc Dis. 2012 Apr;22(4):362-8. doi: 10.1016/j.numecd.2010.07.015. Epub 2010 Dec 24. PMID 21185701
- [Result] van Rompay MI, McKeown NM, Castaneda-Sceppa C, Falcon LM, Ordovas JM, Tucker KL. Acculturation and sociocultural influences on dietary intake and health status among Puerto Rican adults in Massachusetts. J Acad Nutr Diet. 2012 Jan;112(1):64-74. doi: 10.1016/j.jada.2011.08.049. PMID 22389874
- [Result] Perez NA, Weathers B, Willis M, Mendez J. Collaboration across eight research centers: unanticipated benefits and outcomes for project managers. Popul Health Manag. 2013 Feb;16(1):46-52. doi: 10.1089/pop.2012.0024. Epub 2012 Oct 31. PMID 23113631
- [Result] Feng X, Tucker KL, Parnell LD, Shen J, Lee YC, Ordovas JM, Ling WH, Lai CQ. Insulin receptor substrate 1 (IRS1) variants confer risk of diabetes in the Boston Puerto Rican Health Study. Asia Pac J Clin Nutr. 2013;22(1):150-9. doi: 10.6133/apjcn.2013.22.1.09. PMID 23353623
- [Result] Ye X, Scott T, Gao X, Maras JE, Bakun PJ, Tucker KL. Mediterranean diet, healthy eating index 2005, and cognitive function in middle-aged and older Puerto Rican adults. J Acad Nutr Diet. 2013 Feb;113(2):276-81.e1-3. doi: 10.1016/j.jand.2012.10.014. PMID 23351632
- [Result] Moorthy D, Peter I, Scott TM, Parnell LD, Lai CQ, Crott JW, Ordovas JM, Selhub J, Griffith J, Rosenberg IH, Tucker KL, Troen AM. Status of vitamins B-12 and B-6 but not of folate, homocysteine, and the methylenetetrahydrofolate reductase C677T polymorphism are associated with impaired cognition and depression in adults. J Nutr. 2012 Aug;142(8):1554-60. doi: 10.3945/jn.112.161828. Epub 2012 Jun 27. PMID 22739363
- [Result] Ye X, Bhupathiraju SN, Tucker KL. Variety in fruit and vegetable intake and cognitive function in middle-aged and older Puerto Rican adults. Br J Nutr. 2013 Feb 14;109(3):503-10. doi: 10.1017/S0007114512001183. Epub 2012 May 1. PMID 22717056
- [Result] Smith CE, Tucker KL, Lee YC, Lai CQ, Parnell LD, Ordovas JM. Low-density lipoprotein receptor-related protein 1 variant interacts with saturated fatty acids in Puerto Ricans. Obesity (Silver Spring). 2013 Mar;21(3):602-8. doi: 10.1002/oby.20001. PMID 23404896
- [Result] Ma XY, Qiu WQ, Smith CE, Parnell LD, Jiang ZY, Ordovas JM, Tucker KL, Lai CQ. Association between BDNF rs6265 and obesity in the Boston Puerto Rican Health Study. J Obes. 2012;2012:102942. doi: 10.1155/2012/102942. Epub 2012 Dec 27. PMID 23326649
- [Result] Van Rompay MI, McKeown NM, Castaneda-Sceppa C, Ordovas JM, Tucker KL. Carbohydrate nutrition differs by diabetes status and is associated with dyslipidemia in Boston Puerto Rican adults without diabetes. J Nutr. 2013 Feb;143(2):182-8. doi: 10.3945/jn.112.168914. Epub 2012 Dec 26. PMID 23269655
- [Result] Todorova IL, Tucker KL, Jimenez MP, Lincoln AK, Arevalo S, Falcon LM. Determinants of self-rated health and the role of acculturation: implications for health inequalities. Ethn Health. 2013;18(6):563-85. doi: 10.1080/13557858.2013.771147. Epub 2013 Feb 21. PMID 23425383
- [Result] Zheng JS, Arnett DK, Parnell LD, Lee YC, Ma Y, Smith CE, Richardson K, Li D, Borecki IB, Ordovas JM, Tucker KL, Lai CQ. Genetic variants at PSMD3 interact with dietary fat and carbohydrate to modulate insulin resistance. J Nutr. 2013 Mar;143(3):354-61. doi: 10.3945/jn.112.168401. Epub 2013 Jan 9. PMID 23303871
- [Result] Mattei J, Bhupathiraju S, Tucker KL. Higher adherence to a diet score based on American Heart Association recommendations is associated with lower odds of allostatic load and metabolic syndrome in Puerto Rican adults. J Nutr. 2013 Nov;143(11):1753-9. doi: 10.3945/jn.113.180141. Epub 2013 Sep 4. PMID 24005611
- [Result] Zheng JS, Arnett DK, Parnell LD, Smith CE, Li D, Borecki IB, Tucker KL, Ordovas JM, Lai CQ. Modulation by dietary fat and carbohydrate of IRS1 association with type 2 diabetes traits in two populations of different ancestries. Diabetes Care. 2013 Sep;36(9):2621-7. doi: 10.2337/dc12-2607. Epub 2013 Apr 17. PMID 23596181
- [Result] Zheng JS, Arnett DK, Parnell LD, Lee YC, Ma Y, Smith CE, Richardson K, Li D, Borecki IB, Tucker KL, Ordovas JM, Lai CQ. Polyunsaturated Fatty Acids Modulate the Association between PIK3CA-KCNMB3 Genetic Variants and Insulin Resistance. PLoS One. 2013 Jun 27;8(6):e67394. doi: 10.1371/journal.pone.0067394. Print 2013. PMID 23826284
- [Result] Bhupathiraju SN, Lichtenstein AH, Dawson-Hughes B, Hannan MT, Tucker KL. Adherence to the 2006 American Heart Association Diet and Lifestyle Recommendations for cardiovascular disease risk reduction is associated with bone health in older Puerto Ricans. Am J Clin Nutr. 2013 Nov;98(5):1309-16. doi: 10.3945/ajcn.112.056267. Epub 2013 Sep 18. PMID 24047918
- [Result] Smith CE, Tucker KL, Arnett DK, Noel SE, Corella D, Borecki IB, Feitosa MF, Aslibekyan S, Parnell LD, Lai CQ, Lee YC, Ordovas JM. Apolipoprotein A2 polymorphism interacts with intakes of dairy foods to influence body weight in 2 U.S. populations. J Nutr. 2013 Dec;143(12):1865-71. doi: 10.3945/jn.113.179051. Epub 2013 Oct 9. PMID 24108135
- [Result] Jamal-Allial A, Griffith JL, Tucker KL. The longitudinal association of vitamin D serum concentrations & adiposity phenotype. J Steroid Biochem Mol Biol. 2014 Oct;144 Pt A:185-8. doi: 10.1016/j.jsbmb.2013.12.004. Epub 2013 Dec 12. PMID 24333795
- [Result] Zheng JS, Parnell LD, Smith CE, Lee YC, Jamal-Allial A, Ma Y, Li D, Tucker KL, Ordovas JM, Lai CQ. Circulating 25-hydroxyvitamin D, IRS1 variant rs2943641, and insulin resistance: replication of a gene-nutrient interaction in 4 populations of different ancestries. Clin Chem. 2014 Jan;60(1):186-96. doi: 10.1373/clinchem.2013.215251. Epub 2013 Nov 19. PMID 24255076
- [Result] Andrews-Chavez JY, Lee CS, Houser RF, Falcon LM, Tucker KL. Factors associated with alcohol consumption patterns in a Puerto Rican urban cohort. Public Health Nutr. 2015 Feb;18(3):464-73. doi: 10.1017/S1368980014000433. Epub 2014 Apr 8. PMID 24713083
- [Result] Todorova IL, Guzzardo MT, Adams WE, Falcon LM. Gratitude and longing: Meanings of health in aging for Puerto Rican adults in the mainland. J Health Psychol. 2015 Dec;20(12):1602-12. doi: 10.1177/1359105313519155. Epub 2014 Feb 3. PMID 24496056
- [Result] Zheng JS, Lai CQ, Parnell LD, Lee YC, Shen J, Smith CE, Casas-Agustench P, Richardson K, Li D, Noel SE, Tucker KL, Arnett DK, Borecki IB, Ordovas JM. Genome-wide interaction of genotype by erythrocyte n-3 fatty acids contributes to phenotypic variance of diabetes-related traits. BMC Genomics. 2014 Sep 11;15(1):781. doi: 10.1186/1471-2164-15-781. PMID 25213455
- [Result] Arevalo SP, Tucker KL, Falcon LM. Life events trajectories, allostatic load, and the moderating role of age at arrival from Puerto Rico to the US mainland. Soc Sci Med. 2014 Nov;120:301-10. doi: 10.1016/j.socscimed.2014.09.040. Epub 2014 Sep 22. PMID 25265208
- [Result] Berkowitz SA, Gao X, Tucker KL. Food-insecure dietary patterns are associated with poor longitudinal glycemic control in diabetes: results from the Boston Puerto Rican Health study. Diabetes Care. 2014 Sep;37(9):2587-92. doi: 10.2337/dc14-0753. Epub 2014 Jun 26. PMID 24969578
- [Result] Todorova IL, Tejada S, Castaneda-Sceppa C. Perspectives of Puerto Rican Adults about Heart Health and a Potential Community Program. Am J Health Educ. 2014;45(2):76-85. doi: 10.1080/19325037.2013.875961. PMID 26161165
- [Result] Ma Y, Tucker KL, Smith CE, Lee YC, Huang T, Richardson K, Parnell LD, Lai CQ, Young KL, Justice AE, Shao Y, North KE, Ordovas JM. Lipoprotein lipase variants interact with polyunsaturated fatty acids for obesity traits in women: replication in two populations. Nutr Metab Cardiovasc Dis. 2014 Dec;24(12):1323-9. doi: 10.1016/j.numecd.2014.07.003. Epub 2014 Jul 22. PMID 25156894
- [Result] Rodrıguez-Galan MB, Falcon LM. Aging Puerto Ricans' Experiences of Depression Treatment: A New Ethnographic Exploration. Research in the Sociology of Health Care 2014;32:275-303.
- [Result] Adams WE, Todorova ILG, Falcon LM. Puerto Rican Victimization and Crime on the Mainland: The Role of Acculturation. Hisp J Behav Sci. 2015 Feb;37(1):59-74. doi: 10.1177/0739986314564149. Epub 2014 Dec 21. PMID 33223605
- [Result] Flores AM, Nelson J, Martinez Tyson D, Stephenson R, Tucker KL. Physical and functional impairments and physical therapy utilization in cancer survivors of Puerto Rican descent. J Oncol Navigation & Survivorship (JONS-online) 2015;6(3):46-55.
- [Result] Jimenez MP, Osypuk TL, Arevalo S, Tucker KL, Falcon LM. Neighborhood socioeconomic context and change in allostatic load among older Puerto Ricans: The Boston Puerto Rican health study. Health Place. 2015 May;33:1-8. doi: 10.1016/j.healthplace.2015.02.001. Epub 2015 Feb 20. PMID 25706323
- [Result] Adams WE, Todorova IL, Guzzardo MT, Falcon LM. 'The problem here is that they want to solve everything with pills': medication use and identity among Mainland Puerto Ricans. Sociol Health Illn. 2015 Jul;37(6):904-19. doi: 10.1111/1467-9566.12240. Epub 2015 Feb 27. PMID 25720591
- [Result] Arevalo SP, Tucker KL, Falcon LM. Beyond cultural factors to understand immigrant mental health: Neighborhood ethnic density and the moderating role of pre-migration and post-migration factors. Soc Sci Med. 2015 Aug;138:91-100. doi: 10.1016/j.socscimed.2015.05.040. Epub 2015 May 29. PMID 26057720
- [Result] Sotos-Prieto M, Bhupathiraju SN, Falcon LM, Gao X, Tucker KL, Mattei J. A Healthy Lifestyle Score Is Associated with Cardiometabolic and Neuroendocrine Risk Factors among Puerto Rican Adults. J Nutr. 2015 Jul;145(7):1531-40. doi: 10.3945/jn.114.206391. Epub 2015 May 6. PMID 25948783
- [Result] Rioux CL, Tucker KL, Brugge D, Mwamburi M. Medication type modifies inflammatory response to traffic exposure in a population with type 2 diabetes. Environ Pollut. 2015 Jul;202:58-65. doi: 10.1016/j.envpol.2015.03.012. Epub 2015 Mar 24. PMID 25805568
- [Result] Niu J, Sahni S, Liao S, Tucker KL, Dawson-Hughes B, Gao X. Association between Sleep Duration, Insomnia Symptoms and Bone Mineral Density in Older Boston Puerto Rican Adults. PLoS One. 2015 Jul 6;10(7):e0132342. doi: 10.1371/journal.pone.0132342. eCollection 2015. PMID 26147647
- [Result] Palacios C, Trak MA, Betancourt J, Joshipura K, Tucker KL. Validation and reproducibility of a semi-quantitative FFQ as a measure of dietary intake in adults from Puerto Rico. Public Health Nutr. 2015 Oct;18(14):2550-8. doi: 10.1017/S1368980014003218. Epub 2015 Jan 27. PMID 25621587
- [Result] Philip D, Buch A, Moorthy D, Scott TM, Parnell LD, Lai CQ, Ordovas JM, Selhub J, Rosenberg IH, Tucker KL, Troen AM. Dihydrofolate reductase 19-bp deletion polymorphism modifies the association of folate status with memory in a cross-sectional multi-ethnic study of adults. Am J Clin Nutr. 2015 Nov;102(5):1279-88. doi: 10.3945/ajcn.115.111054. Epub 2015 Sep 9. PMID 26354538
- [Result] Dashti HS, Aslibekyan S, Scheer FA, Smith CE, Lamon-Fava S, Jacques P, Lai CQ, Tucker KL, Arnett DK, Ordovas JM. Clock Genes Explain a Large Proportion of Phenotypic Variance in Systolic Blood Pressure and This Control Is Not Modified by Environmental Temperature. Am J Hypertens. 2016 Jan;29(1):132-40. doi: 10.1093/ajh/hpv082. Epub 2015 Jun 4. PMID 26045533
- [Result] Guzzardo MT, Todorova IL, Adams WE, Falcón LM. "Half Here, Half There": Dialogical Selves Among Older Puerto Ricans of the Diaspora. J Constr Psychol 2016;29(1):51-65.
- [Result] Guzzardo MT, Adams WE, Todorova IL, Falcón LM. Resonating sentiments on Puerto Rican identity through poetry: Voices of the diaspora. Qualitative Inquiry 2016 doi: 10.1177/1077800415622485
- [Result] Sotos-Prieto M, Bhupathiraju SN, Falcon LM, Gao X, Tucker KL, Mattei J. Association between a Healthy Lifestyle Score and inflammatory markers among Puerto Rican adults. Nutr Metab Cardiovasc Dis. 2016 Mar;26(3):178-84. doi: 10.1016/j.numecd.2015.12.004. Epub 2015 Dec 29. PMID 26838054
- [Result] Bigornia SJ, Lichtenstein AH, Harris WS, Tucker KL. Associations of erythrocyte fatty acid patterns with insulin resistance. Am J Clin Nutr. 2016 Mar;103(3):902-9. doi: 10.3945/ajcn.115.123604. Epub 2016 Feb 10. PMID 26864364
- [Result] Bigornia SJ, Harris WS, Falcon LM, Ordovas JM, Lai CQ, Tucker KL. The Omega-3 Index Is Inversely Associated with Depressive Symptoms among Individuals with Elevated Oxidative Stress Biomarkers. J Nutr. 2016 Apr;146(4):758-66. doi: 10.3945/jn.115.222562. Epub 2016 Mar 2. PMID 26936135
- [Result] Blanco-Rojo R, Delgado-Lista J, Lee YC, Lai CQ, Perez-Martinez P, Rangel-Zuniga O, Smith CE, Hidalgo B, Alcala-Diaz JF, Gomez-Delgado F, Parnell LD, Arnett DK, Tucker KL, Lopez-Miranda J, Ordovas JM. Interaction of an S100A9 gene variant with saturated fat and carbohydrates to modulate insulin resistance in 3 populations of different ancestries. Am J Clin Nutr. 2016 Aug;104(2):508-17. doi: 10.3945/ajcn.116.130898. Epub 2016 Jul 20. PMID 27440084
- [Result] Mattei J, Mendez J, Falcon LM, Tucker KL. Perceptions and Motivations to Prevent Heart Disease among Puerto Ricans. Am J Health Behav. 2016 May;40(3):322-31. doi: 10.5993/AJHB.40.3.4. PMID 27103411
- [Result] Wong JC, Scott T, Wilde P, Li YG, Tucker KL, Gao X. Food Insecurity Is Associated with Subsequent Cognitive Decline in the Boston Puerto Rican Health Study. J Nutr. 2016 Sep;146(9):1740-5. doi: 10.3945/jn.115.228700. Epub 2016 Jul 27. PMID 27466603
- [Result] Smith CE, Coltell O, Sorli JV, Estruch R, Martinez-Gonzalez MA, Salas-Salvado J, Fito M, Aros F, Dashti HS, Lai CQ, Miro L, Serra-Majem L, Gomez-Gracia E, Fiol M, Ros E, Aslibekyan S, Hidalgo B, Neuhouser ML, Di C, Tucker KL, Arnett DK, Ordovas JM, Corella D. Associations of the MCM6-rs3754686 proxy for milk intake in Mediterranean and American populations with cardiovascular biomarkers, disease and mortality: Mendelian randomization. Sci Rep. 2016 Sep 14;6:33188. doi: 10.1038/srep33188. PMID 27624874
- [Result] Noel SE, Arevalo S, Smith CE, Lai CQ, Dawson-Hughes B, Ordovas JM, Tucker KL. Genetic admixture and body composition in Puerto Rican adults from the Boston Puerto Rican Osteoporosis Study. J Bone Miner Metab. 2017 Jul;35(4):448-455. doi: 10.1007/s00774-016-0775-6. Epub 2016 Sep 14. PMID 27628044
- [Result] Smith CE, Fullerton SM, Dookeran KA, Hampel H, Tin A, Maruthur NM, Schisler JC, Henderson JA, Tucker KL, Ordovas JM. Using Genetic Technologies To Reduce, Rather Than Widen, Health Disparities. Health Aff (Millwood). 2016 Aug 1;35(8):1367-73. doi: 10.1377/hlthaff.2015.1476. PMID 27503959
- [Result] Zhang Y, Cifuentes M, Gao X, Amaral G, Tucker KL. Age- and gender-specific associations between insomnia and falls in Boston Puerto Rican adults. Qual Life Res. 2017 Jan;26(1):25-34. doi: 10.1007/s11136-016-1374-7. Epub 2016 Jul 23. PMID 27448438
- [Result] Mattei J, Sotos-Prieto M, Bigornia SJ, Noel SE, Tucker KL. The Mediterranean Diet Score Is More Strongly Associated with Favorable Cardiometabolic Risk Factors over 2 Years Than Other Diet Quality Indexes in Puerto Rican Adults. J Nutr. 2017 Apr;147(4):661-669. doi: 10.3945/jn.116.245431. Epub 2017 Mar 8. PMID 28275099
- [Derived] Dinesh D, Morgan XC, Kim H, Scott TM, Garelnabi M, Lee JS, Mangano KM, Nguyen LH, Huttenhower C, Tucker KL, Palacios N. Gut Microbial Variations Associated With Proton Pump Inhibitor Use in the Boston Puerto Rican Health Study. Pharmacol Res Perspect. 2026 Feb;14(1):e70205. doi: 10.1002/prp2.70205. PMID 41437205
- [Derived] Dinesh D, Lee JS, Scott TM, Tucker KL, Palacios N. Bowel Health, Laxative Use, and Cognitive Function in Older Puerto Rican Adults. J Aging Res. 2025 Jul 24;2025:2674457. doi: 10.1155/jare/2674457. eCollection 2025. PMID 40746372
- [Derived] Guan Y, Ebrahimzadeh SA, Cheng CH, Chen W, Leung T, Bigornia S, Palacios N, Garelnabi MO, Scott T, Bhadelia R, Tucker KL, Koo BB; Alzheimer's Disease Neuroimaging Initiative. Association of Diabetes and Hypertension With Brain Structural Integrity and Cognition in the Boston Puerto Rican Health Study Cohort. Neurology. 2022 Apr 12;98(15):e1534-e1544. doi: 10.1212/WNL.0000000000200120. Epub 2022 Mar 30. PMID 35354581
- [Derived] Flores AC, Heron C, Kim JI, Martin B, Al-Shaar L, Tucker KL, Gao X. Prospective Study of Plant-Based Dietary Patterns and Diabetes in Puerto Rican Adults. J Nutr. 2021 Dec 3;151(12):3795-3800. doi: 10.1093/jn/nxab301. PMID 34515303
- [Derived] Mangano KM, Noel SE, Lai CQ, Christensen JJ, Ordovas JM, Dawson-Hughes B, Tucker KL, Parnell LD. Diet-derived fruit and vegetable metabolites show sex-specific inverse relationships to osteoporosis status. Bone. 2021 Mar;144:115780. doi: 10.1016/j.bone.2020.115780. Epub 2020 Dec 2. PMID 33278656
- [Derived] Mangano KM, Noel SE, Sahni S, Tucker KL. Higher Dairy Intakes Are Associated with Higher Bone Mineral Density among Adults with Sufficient Vitamin D Status: Results from the Boston Puerto Rican Osteoporosis Study. J Nutr. 2019 Jan 1;149(1):139-148. doi: 10.1093/jn/nxy234. PMID 30601986
- [Derived] Mattei J, McClain AC, Falcon LM, Noel SE, Tucker KL. Dietary Acculturation among Puerto Rican Adults Varies by Acculturation Construct and Dietary Measure. J Nutr. 2018 Nov 1;148(11):1804-1813. doi: 10.1093/jn/nxy174. PMID 30383277
- [Derived] Bhupathiraju SN, Dawson-Hughes B, Hannan MT, Lichtenstein AH, Tucker KL. Centrally located body fat is associated with lower bone mineral density in older Puerto Rican adults. Am J Clin Nutr. 2011 Oct;94(4):1063-70. doi: 10.3945/ajcn.111.016030. Epub 2011 Aug 24. PMID 21865328